CLINICAL TRIAL: NCT01486056
Title: ECG Vector Determination for Model 106 Generator Implant Site Selection
Brief Title: ECG Vector Determination
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E-35
Record Dates: First submitted 2011-11-28; First posted 2011-12-06 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Epilepsy
Keywords: epilepsy; ECG; device placement
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy patients, may have epilepsy: Subjects at least 12 years old and in general good health for Phase I, and at least 18 years old and in general good health for Phase II. It is desired, but not required, for subjects to have epilepsy and taking at least 1 antiepileptic medication.

SUMMARY:
This is a prospective, unblinded, non-randomized, descriptive study designed to collect ECG data.

DETAILED DESCRIPTION:
This is a prospective, unblinded, non-randomized, descriptive study designed to collect ECG data and determine the process for proper generator and lead placement. The study will be conducted in two phases: Phase I includes ECG data collection from human subjects; Phase II, the Implant Instructions for Use will be evaluated by Cyberonics' Clinical Engineers based on the activities of five to eight experienced VNS surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. At least 12 years old and in general good health for Phase I. At least 18 years old and in general good health for Phase II.
2. Patients or their guardians must be willing to provide signed informed consent/assent and HIPAA authorization. Note: Patients diagnosed with epilepsy and taking at least 1 antiepileptic medication are desired but not required for the study.

Exclusion Criteria:

1. History of pathologically significant cardiac arrhythmias including but not limited to atrial fibrillation or flutter, chronotropic incompetence, supraventricular tachycardia, ventricular flutter or fibrillation, or implantation of a permanent cardiac pacemaker or defibrillator.
2. Currently present existing signs of skin irritation or rash on the left neck or upper left chest as determined by the PI.
3. History of physical adverse reaction to adhesive electrodes.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects 12 years and older in general good health, preferably with epilepsy and on at least 1 antiepileptic medication.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To correlate ECG amplitude with prospective VNS implant sites. | up to 2 days
  This study is designed to collect ECG data to determine the process for proper generator and lead placement.

SECONDARY OUTCOMES:
To identify potential VNS implant sites associated with low ECG amplitudes. | up to 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Denham, DO, Principal Investigator — Clinical Trails of Texas, Inc.; Bryan Olin, Ph.D, Study Director — Cyberonics, Inc.
Locations (1):
- Clinical Trials of Texas, Inc., San Antonio, Texas, United States

REFERENCES:
- [Background] VAN BUREN JM. Some autonomic concomitants of ictal automatism; a study of temporal lobe attacks. Brain. 1958 Dec;81(4):505-28. doi: 10.1093/brain/81.4.505. No abstract available. PMID 13618449
- [Background] Marshall DW, Westmoreland BF, Sharbrough FW. Ictal tachycardia during temporal lobe seizures. Mayo Clin Proc. 1983 Jul;58(7):443-6. PMID 6865478
- [Background] Keilson MJ, Hauser WA, Magrill JP. Electrocardiographic changes during electrographic seizures. Arch Neurol. 1989 Nov;46(11):1169-70. doi: 10.1001/archneur.1989.00520470023018. PMID 2818251
- [Background] Smith PE, Howell SJ, Owen L, Blumhardt LD. Profiles of instant heart rate during partial seizures. Electroencephalogr Clin Neurophysiol. 1989 Mar;72(3):207-17. doi: 10.1016/0013-4694(89)90245-9. PMID 2465123
- [Background] O'Donovan C, Burgess R, Luders H., Computerized seizure detection based on heart rate changes. Epilepsia 1995;36(suppl 4):7.
- [Background] Schernthaner C, Lindinger G, Potzelberger K, Zeiler K, Baumgartner C. Autonomic epilepsy--the influence of epileptic discharges on heart rate and rhythm. Wien Klin Wochenschr. 1999 May 21;111(10):392-401. PMID 10413832
- [Background] Leutmezer F, Schernthaner C, Lurger S, Potzelberger K, Baumgartner C. Electrocardiographic changes at the onset of epileptic seizures. Epilepsia. 2003 Mar;44(3):348-54. doi: 10.1046/j.1528-1157.2003.34702.x. PMID 12614390
- [Background] Di Gennaro G, Quarato PP, Sebastiano F, Esposito V, Onorati P, Grammaldo LG, Meldolesi GN, Mascia A, Falco C, Scoppetta C, Eusebi F, Manfredi M, Cantore G. Ictal heart rate increase precedes EEG discharge in drug-resistant mesial temporal lobe seizures. Clin Neurophysiol. 2004 May;115(5):1169-77. doi: 10.1016/j.clinph.2003.12.016. PMID 15066542